CLINICAL TRIAL: NCT07364305
Title: HAIC Combined With Immune Therapy for Advanced, Non-Resectable ICC: A Single-Arm, Multicenter Phase II Clinical Trial
Brief Title: HAIC Combined With Immune Therapy for Advanced, Non-Resectable ICC
Acronym: Lalo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Chengjun Sui,MD, Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lalo; 20241130 (Other Grant/Funding Number: Shanghai Municipal Health Commission)
Record Dates: First submitted 2026-01-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: ICC; Advanced Cancer
Keywords: HAIC; Immunotherapy
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC combined with PD-L1 inhibitor (Experimental): Hepatic arterial infusion chemotherapy (HAIC) combined with PD-L1 inhibitor 1.Therapy:hepatic
  arterial infusion chemotherapy (HAIC) hepatic arterial infusion chemotherapy (HAIC) : GemCis regimen was
  adopted, with the specific regimen as follows: Cisplatin 20mg/m2, maintained for 3 hours. Gemcitabine 0.6g/m2,
  maintained for 1 hour , repeated once every 3 weeks, and 4-6 cycles of treatment (the specific number of cycles
  was determined by the investigator according to the patient's condition). 2. PD-L1 inhibitor Drug: Durvalumab
  OR pembrolizumab Durvalumab: During combination therapy: 1500 mg, Q3W, during combination therapy, on days 3-5
  of each 3-week cycle (determined by the investigator); during maintenance therapy: 1500 mg Q4W Pembrolizumab:
  During combination therapy: 200 mg, Q3W, during combination therapy, on days 3-5 of each 3-week cycle
  (determined by the investigator); during maintenance therapy: 200 mg Q4W
  Interventions: Drug: PD-L1 inhibitor; Procedure: HAIC

INTERVENTIONS:
Drug: PD-L1 inhibitor — PD-L1 inhibitor Drug: Durvalumab OR pembrolizumab Durvalumab: During combination therapy: 1500 mg, Q3W, during combination therapy, on days 3-5 of each 3-week cycle (determined by the investigator); during maintenance therapy: 1500 mg Q4W Pembrolizumab: During combination therapy: 200 mg, Q3W, during combination therapy, on days 3-5 of each 3-week cycle (determined by the investigator); during maintenance therapy: 200 mg Q4W
Procedure: HAIC — Hepatic arterial infusion chemotherapy (HAIC) combined with PD-L1 inhibitor 1.Therapy:hepatic arterial infusion chemotherapy (HAIC) hepatic arterial infusion chemotherapy (HAIC) : GemCis regimen was adopted, with the specific regimen as follows: Cisplatin 20mg/m2, maintained for 3 hours. Gemcitabine 0.6g/m2, maintained for 1 hour , repeated once every 3 weeks, and 4-6 cycles of treatment (the specific number of cycles was determined by the investigator according to the patient's condition).

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) has a poor prognosis. The aim of this study is to investigate the efficacy and safety of GP-HAIC combined with immunosuppressants in the treatment of initially unresectable ICC patients, as well as its role in conversion therapy. A prospective study was conducted on the data of locally advanced unresectable ICC patients receiving GC-HAIC combined with immunosuppressive therapy, evaluating the treatment efficacy and safety.

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC)-GC（Gemcitabine+Cisplatin） combined with Durvalumab OR Pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

1. Age: Age ≥ 18 years old.
2. Diagnosis: Advanced unresectable intrahepatic cholangiocarcinoma (ICC) diagnosed by histology or imaging.
3. Measurable lesion: At least one measurable tumor lesion (according to RECIST 1.1 criteria).
4. Physical fitness status: The Eastern Cancer Collaboration Group (ECOG) physical fitness status score is 0 or 1.
5. Expected lifespan: Expected lifespan ≥ 3 months.
6. Liver function: Child Pugh classification A or B.
7. Organ function: It has sufficient organ function and laboratory tests meet the requirements of the protocol.
8. Not receiving relevant treatment: Not receiving systematic treatment for ICC.

Exclusion Criteria:

1. Previous treatment: Previously received systemic treatment for ICC.
2. Poor physical condition: ECOG physical condition score ≥ 2.
3. Poor liver function: Child Pugh grading>8.
4. Short life expectancy: Life expectancy is less than 3 months.
5. Merge with other malignant tumors: have other malignant tumors or a history of other malignant tumors.
6. Serious organ dysfunction: There is severe dysfunction in organs such as the heart, brain, lungs, and kidneys.
7. Drug allergy or intolerance: Allergic to the investigational drug or its excipients.
8. Other: Other situations that the researcher deems unsuitable to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 year
  Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR was defined as 2 CRs or 2 PRs with no evidence of progression in-between. Patients who discontinued randomized treatment without progression, received a subsequent anti-cancer therapy and then responded were not included as responders for ORR.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Overall Survival (OS) was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Progression-free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS based on investigator assessments according to RECIST version 1.1 was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was calculated using the Kaplan-Meier technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No